CLINICAL TRIAL: NCT01559402
Title: Application of Protective Ventilation Improves Oxygenation During and After Anesthesia. Is it Possible That a Special Procedure, an Oxygenation Test, Can Replace Arterial Blood Gases When Evaluating Oxygenation?
Brief Title: Oxygenation Test During General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Västmanland (Other)
Responsible Party: Principal Investigator, Lennart Edmark, Principal Investigator, Region Västmanland
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: Dnr 2011 / 462
Record Dates: First submitted 2012-03-12; First posted 2012-03-21 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-08

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid | interventions — Oxygen; AIEOP acute lymphoblastic leukemia protocol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Start O2 100% and CPAP 10, end O2 100%. (Experimental): This arm describes some aspects of ventilation during anesthesia for laparoscopic gastric bypass. Pre-oxygenation is with an inspiratory oxygen fraction(FIO2) of 1.0, supplied by a continuous positive airway pressure of 10 centimeters of water(cmH2O), during anesthesia a positive end-expiratory pressure of 10 cmH2O is used and during emergence from anesthesia a FIO2 of 1.0 is used. The intervention associated with this arm is labeled CPAP and 100% oxygen.
  Interventions: Procedure: CPAP and 100% oxygen
- Start O2 100% and CPAP 10, end O2 31%. (Experimental): This arm describes some aspects of ventilation during anesthesia for laparoscopic gastric bypass. Pre-oxygenation is with a FIO2 of 1.0, supplied by a continuous positive airway pressure of 10 cmH2O, during anesthesia a positive end-expiratory pressure of 10 cmH2O is used and during emergence from anesthesia a FIO2 of 0.3 is used. The intervention associated with this arm is labeled CPAP and 31% oxygen.
  Interventions: Procedure: CPAP and 31% oxygen
- Start O2 100% and CPAP 0, end O2 100%. (Experimental): This arm describes some aspects of ventilation during anesthesia for laparoscopic gastric bypass. Pre-oxygenation is with a FIO2 of 1.0, without a continuous positive airway pressure, during anesthesia a positive end-expiratory pressure of 10 cmH2O is used and during emergence from anesthesia a FIO2 of 1.0 is used. The intervention associated with this arm is labeled No CPAP and 100% oxygen.
  Interventions: Procedure: No CPAP and 100% oxygen

INTERVENTIONS:
Procedure: CPAP and 100% oxygen — During pre oxygenation and induction of anesthesia 100 % oxygen is used with a continuous positive airway pressure of 10 cmH2O, during maintenance of anesthesia a positive endexpiratory pressure of 10 cm H20 is used with controlled volume ventilation aiming at an end tidal carbon dioxide (CO2) level of 5 %. During emergence from anesthesia 100 % oxygen is used.
  Other Names: Preventive ventilation
  Arms: Start O2 100% and CPAP 10, end O2 100%.
Procedure: CPAP and 31% oxygen — During pre oxygenation and induction of anesthesia 100 % oxygen is used with a continuous positive airway pressure of 10 cm H2O, during maintenance of anesthesia a positive endexpiratory pressure of 10 cm H20 is used with controlled volume ventilation aiming at an end tidal CO2 level of 5 %. During emergence from anesthesia 31 % inspiratory oxygen or the inspiratory oxygen level needed to achieve a SpO2 of at least 96 % (if 31 % oxygen is not enough), is used.
  Other Names: Preventive ventilation
  Arms: Start O2 100% and CPAP 10, end O2 31%.
Procedure: No CPAP and 100% oxygen — This intervention follows a standard protocol without the use CPAP during induction of anesthesia.
  Other Names: Standard protocol.
  Arms: Start O2 100% and CPAP 0, end O2 100%.

SUMMARY:
The study investigates if applying a special ventilatory strategy during anesthesia for laparoscopic gastric by pass, produces less atelectasis and better oxygenation in spite of using 100 % oxygen during pre oxygenation and induction of anesthesia. The study investigates oxygenation with blood gas samples but also with a new method that might give more information without the use of blood gas samples.

Primary: Oxygenation in patients with morbid obesity improves if preoxygenation, induction and maintenance of anesthesia is performed with either a continuous positive airway pressure (CPAP) or a positive end expiratory pressure (PEEP), respectively, of 10 cm H2O, in comparison to a technique without CPAP but with a PEEP of 10 cm H2O.

Secondary: The improved oxygenation during anesthesia can be prolonged inte the postoperative period if emergence from anesthesia is performed without high levels of oxygen.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients scheduled for elective surgery of Morbid Obesity.
* ASA 1-2. (ASA = American Society of Anesthesiologists classification).
* "Body mass index" (BMI) ≥ 35 but < 50

Exclusion Criteria:

* "ASA 3"
* Anticipated difficult intubation.
* Major bleeding.
* Problems with ventilation necessitating protocol aberrations.
* Obstructive sleep apnea syndrome with CPAP treatment at home.
* Angina Pectoris

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change in peripheral O2 saturation(SpO2)during and 1 hour after anesthesia in comparison to awake before anesthesia. | Change in SpO2 from 5 min before start of anesthesia, to 5 min after intubation, 5 min before extubation and 1 hour after extubation.
  During anesthesia SpO2 is measured at three different levels of oxygen; 21, 26 and 31 % respectively as long as SpO2 does not go lower than 87 % and compared to SpO2 immediately before anesthesia. SpO2 breathing air one hour after anesthesia is compared to SpO2 before anesthesia.

SECONDARY OUTCOMES:
Arterial blood gas values for saturation (SaO2) | 5 min before anesthesia, 5 min after intubation, 5 min before extubation and 1 hour after anesthesia.
  During anesthesia SaO2 is measured at three different levels of oxygen; 21, 26 and 31 % respectively as long as SpO2 (sic! does not go lower than 87 % and compared to SaO2 immediately before anesthesia. SaO2 breathing air one hour after anesthesia is compared to SaO2 before anesthesia.
Arterial oxygen tension (PaO2) | 5 min before start of anesthesia, 5 min after intubation, 5 min before extubation and 1 hour after extubation.
  During anesthesia PaO2 is measured at three different levels of oxygen; 21, 26 and 31 % respectively as long as SpO2 (sic) does not go lower than 87 % and compared to PaO2 immediately before anesthesia. PaO2 breathing air one hour after anesthesia is compared to PaO2 before anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Göran Hedenstierna, Prof., Principal Investigator — Uppsala University Hospital
Locations (1):
- Operationskliniken, Västmanlands sjukhus Västerås, Västerås, Sweden